CLINICAL TRIAL: NCT02156687
Title: A Prospective Randomized Trial Comparing Restorelle Y Mesh vs. Restorelle Dual Flat Mesh for Laparoscopic and Robotic-assisted Laparoscopic Sacrocolpopexy
Brief Title: Randomized Trial of Y Mesh vs Dual Mesh
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 14-354
Record Dates: First submitted 2014-06-02; First posted 2014-06-05 (Estimated); Results first posted 2020-10-29 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Prolapse
MeSH Terms: conditions — Prolapse

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cololast, Inc. Restorell Y mesh (Active Comparator): Y mesh
  Interventions: Device: Y mesh
- Coloplast, Inc. Restorelle Dual flat mesh (Active Comparator): Dual flat mesh
  Interventions: Device: Dual flat mesh

INTERVENTIONS:
Device: Y mesh — Y mesh
  Other Names: Cololast, Inc. Restorell Y mesh
  Arms: Cololast, Inc. Restorell Y mesh
Device: Dual flat mesh — Dual flat mesh
  Other Names: Coloplast, Inc. Restorelle Dual flat mesh
  Arms: Coloplast, Inc. Restorelle Dual flat mesh

SUMMARY:
The primary objective of the proposed study is to determine the difference in suturing time when using the restorelle Y mesh versus the restorelle dual flat mesh at the time of laparoscopic and robotic-assisted laparoscopic sacrocolpopexy.

Hypothesis: Suturing time when using the restorelle Y mesh will be faster than when using the restorelle dual flat mesh at the time of laparoscopic and robotic-assisted laparoscopic sacrocolpopexy.

DETAILED DESCRIPTION:
Study Design: Randomized single-blind prospective clinical trial

Primary Outcomes:

1. Total Suturing time for mesh placement = time from insertion of Y mesh or first flat mesh arm into pelvis to last sacral suture placed
2. Total Case time = Incision to end of closure

Secondary Outcomes:

Post-operative patient outcomes at 24-months

* Pelvic Floor Dysfunction Inventory (PFDI-20)
* Pelvic Organ Prolapse Distress Inventory (POPDI)
* Colorectal Anal Distress Inventory (CRADI)
* Urogenital Distress Inventory (UDI)
* Objective Recurrence (POP-Q)
* Subjective Recurrence (vaginal bulge)
* Reported mesh erosion

Study Population: Study subjects will be recruited from patients that present to the Center of Urogynecology and Pelvic Floor Disorders in the Department of Obstetrics and Gynecology at the Cleveland Clinic main campus, Hillcrest Hospital and Fairview Hospital, and their surgeries will be performed at either one of these sites.

Study Procedures:

Study Identification and Recruitment Potential subjects will be identified by members of the Center for Urogynecology and Pelvic Reconstructive Surgery at the Cleveland Clinic main campus and Fairview Hospital. Eligible patients that agree to participate will be provided written informed consent administered by the collaborators listed on this Investigational Research Board (IRB) proposal at Cleveland Clinic Main campus and Fairview Hospitals.

Randomization All subjects will be predetermined by their surgeon to undergo either a laparoscopic or robotic assisted laparoscopic sacrocolpopexy depending upon their clinical evaluation. The participants will then be randomized to either Y mesh or dual flat mesh sacrocolpopexy according to a computer-generated randomization schedule with random block sizes with the use of the SAS statistical software package (SAS Institute, Cary, NC). Randomization will be carried out by provider. All patients will be blinded to their assignment.

Office Interventions In addition to a standardized evaluation including the history and physical examination, patients will be asked to complete the Pelvic Floor Distress Inventory (PFDI-20) questionnaire at the pre-operative visit as well as the 6, 12 and 24-month postoperative visit. Completion of these questionnaire is the only additional assessment that is specific to participation in this study and is not usually included as part of the standard care of sacrocolpopexy. It should take no more than 10-15 minutes to complete the questionnaire. The study subjects will not be exposed to any additional risk by participating in this study except for the inconvenience of completing the questionnaire.

Surgical Interventions Laparoscopic sacrocolpopexy will be performed using four ports: an umbilical port for the laparoscope, two ports (either 5 or 10/12 mm) in the bilateral lower quadrants, and one 5-mm port placed at the level of the umbilicus, lateral to the rectus muscle on either side for retraction. The robotic-assisted hysterectomy will be performed using the da Vinci Surgical System (Intuitive Surgical Inc., Sunnyvale, CA, USA) using five ports: a 12mm umbilical port for the laparoscopic, two 8 mm robotic ports placed 2cm inferior and 9-10cm lateral to the umbilicus bilaterally, an 8mm robotic port placed in the left axillary line at the level of the umbilicus, and a 8mm or 10/12mm accessory port either in the right upper quadrant approximately 3cm distal from the costal margin, or in the right lower quadrant, 2cm above and medial to the anterior superior iliac spine.

If a supracervical hysterectomy is to be performed, it will be done in a standard fashion. A uterine manipulator will be placed inside of the uterus. The round ligaments will be transected using cautery. The fallopian tubes and ovaries will be left in situ or removed at the time of hysterectomy depending upon the preoperative decision made between the surgeon and patient. The uterine arteries and cardinal ligaments will be cauterized laparoscopically. The uterus will be amputated at the level of the internal cervical os and the endocervical canal will be cauterized.

The sacrocolpopexy will also be performed and in a standard fashion. An end-to-end anastomosis (EEA) sizer will be placed in the vagina for manipulation of the apex as well as in the rectum for delineation of the rectovaginal septum. First, the presacral dissection will be performed with a longitudinal peritoneal incision over the sacral promontory and there is identification of the anterior longitudinal ligament. Dissection is then done caudally through the peritoneum and subperitoneal fat down to the level of the posterior cul-de-sac. The vagina is elevated cephalad using the EEA sizer and the peritoneum overlying the anterior vaginal apex is incised transversely, and the bladder is dissected off the anterior vagina using sharp dissection, creating a 4 to 5 cm pocket. If this plane is difficult to establish, the bladder will be filled in a retrograde fashion to find the correct dissection plane. Similarly, the peritoneum overlying the posterior vagina is incised, and dissection is then done overlying the vagina and extending into the posterior cul-de-sac, creating a 4 to 5 cm pocket. Once dissection is complete, the mesh graft is prepared. Subjects will have been randomized to either one of two mesh grafts:

1. Restorelle Y mesh

   * The mesh is introduced into the pelvis through one of the ports.
   * First, either then anterior or the posterior arm is fixed to the anterior or posterior vaginal wall using 5 delayed- absorbable (PDS) No. 2-0 sutures in an interrupted fashion, 1 to 2 cm apart from each other.
   * The opposing arm of the graft is then attached to either the anterior or posterior vaginal wall, depending on which arm was placed first, in a similar fashion using 5 delayed- absorbable (PDS) No. 2-0 sutures in an interrupted fashion, 1 to 2 cm apart from each other.
   * The stem portion of the graft is then brought to the sacral promontory and sutured to the anterior longitudinal ligament using 2 permanent (prolene) No. 0 sutures. The excess mesh is then trimmed.
2. Restorelle dual flat mesh: 2 pieces of 15 x 4 cm mesh

   * One mesh arm is introduced into the pelvis through one of the ports.
   * The arm is fixed to the anterior or posterior vaginal wall using 5 delayed- absorbable (PDS) No. 2-0 sutures in an interrupted fashion, 1 to 2 cm apart from each other.
   * The second mesh arm is then introduced into the pelvis through one of the ports.
   * The arm is fixed to either the anterior or posterior vaginal wall, depending on where the first arm was placed, using 5 delayed- absorbable (PDS) No. 2-0 sutures in an interrupted fashion, 1 to 2 cm apart from each other.
   * The two arms are then brought to the sacral promontory and sutured together to the anterior longitudinal ligament using 2 permanent (prolene) No. 0 sutures. The excess mesh is then trimmed.

The peritoneum is then closed over the exposed graft with absorbable suture. Routine cystoscopy will also be performed in order to assess for lower urinary tract injury. A vaginal exam is performed, and an anterior and/or posterior colporrhaphy and perineorrhaphy are performed if needed. Anti-incontinence procedures may also be performed if needed.

**In laparoscopic cases, all suturing will be done extracorporeally while intracorporeal knot-tying technique will be performed in robot assisted laparoscopic cases.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18, who are to undergo laparoscopic or robotic laparoscopic sacrocolpopexy for pelvic organ prolapse
* Other concomitant laparoscopic or prolapse and anti-incontinence procedures (e.g., laparoscopic supracervical hysterectomy, cystocele repair, rectocele repair or mid-urethral sling procedures) will be performed at the primary surgeon's discretion.

Exclusion Criteria:

* Inability to comprehend written and/or spoken English
* Inability to provide informed consent
* Medical illness precluding laparoscopy
* Need for concomitant surgeries not related to pelvic organ prolapse or incontinence
* Sacrocolpoperineopexy

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2014-04-14 (Actual); Primary Completion 2019-11-07 (Actual); Study Completion 2020-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cecile Unger, M.D., Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Coloplast, Inc. Restorelle Y Mesh: Subjects implanted with Coloplast, Inc. Restorelle Y mesh at the time of minimally invasive sacrocolpopexy.
- Coloplast, Inc. Restorelle Dual Flat Mesh: Subjects implanted with Coloplast, Inc. Restorelle Dual flat mesh at the time of minimally invasive sacrocolpopexy.
Period: Overall Study
Arm/Group | Coloplast, Inc. Restorelle Y Mesh | Coloplast, Inc. Restorelle Dual Flat Mesh
Started | 30 | 29
Completed | 20 | 24
Not Completed | 10 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cololast, Inc. Restorell Y Mesh | Coloplast, Inc. Restorelle Dual Flat Mesh | Total
Number analyzed (Participants) | 30 | 29 | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.3 (7.3) | 62.4 (8.1) | 61 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 29 | 59
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 28 | 27 | 55
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 28.9 (3.5) | 28.2 (4.2) | 28.5 (3.9)
Tobacco use [Count of Participants; unit: Participants] | 2 | 3 | 5
Parity [Median (Full Range); unit: pregnancies] | 3 [1 to 6] | 2 [1 to 10] | 3 [1 to 6]
Prior prolapse surgery [Count of Participants; unit: Participants] | 15 | 15 | 30
Prolapse Stage 1 [Count of Participants; unit: Participants] — Patients who had Prolapse stage 1 based on POP-Q exam; this is a standardized measure. The most distal portion of the prolapse is >1 cm above the level of the hymen (i.e., its quantitation value is <-1 cm). Very mild prolapse - organs are still fairly well supported by the pelvic floor.
  Participants | 0 | 0 | 0
Prolapse Stage 2 [Count of Participants; unit: Participants] — Patients who had Prolapse stage 2 based on POP-Q exam; this is a standardized measure. The most distal portion of the prolapse is ≤1 cm proximal to or distal to the plane of the hymen (i.e., its quantitation value is ≥-1 cm but ≤+1 cm). Pelvic floor organs have begun to fall, but are still contained inside the vagina.
  Participants | 9 | 10 | 19
Prolapse Stage 3 [Count of Participants; unit: Participants] — Patients who had Prolapse stage 3 based on POP-Q exam; this is a standardized measure. The most distal portion of the prolapse is >1 cm below the plane of the hymen but protrudes no further than 2 cm less than the total vaginal length in centimeters (i.e., its quantitation value is >+1 cm but <+[TVL-2] cm). Pelvic floor organs have fallen to, or beyond the opening of the vagina.
  Participants | 20 | 17 | 37
Prolapse Stage 4 [Count of Participants; unit: Participants] — Patients who had Prolapse stage 4 based on POP-Q exam; this is a standardized measure. Essentially, complete eversion of the total length of the lower genital tract is demonstrated. The distal portion of the prolapse protrudes to at least (TVL-2) cm (i.e., its quantitation value is ≥+[TVL-2] cm). In most instances, the leading edge of stage IV prolapse is the cervix or vaginal cuff scar. Pelvic floor organs have fallen completely through the vaginal opening.
  Participants | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Total Suturing Time for Mesh Placement = Time From Insertion of Y Mesh or First Flat Mesh Arm Into Pelvis to Last Sacral Suture Placed
Time Frame: one day intraoperative
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- Coloplast, Inc. Restorelle Y Mesh: Y mesh
  Y mesh: Y mesh
Arm/Group | Coloplast, Inc. Restorelle Y Mesh | Coloplast, Inc. Restorelle Dual Flat Mesh
Number analyzed (Participants) | 30 | 29
minutes | 46 (14.7) | 46.3 (12.3)

2. Primary Outcome: Total OR Time = Operating Room Time of Entry and Exit
Time Frame: one day intraoperative
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Coloplast, Inc. Restorelle Y Mesh | Coloplast, Inc. Restorelle Dual Flat Mesh
Number analyzed (Participants) | 30 | 29
minutes | 204.2 (52.8) | 204.5 (43.7)

3. Secondary Outcome: Post-operative Mean Difference POPDI at 24 Months
Description: Mean difference between baseline (pre-procedure) and 24-months post-procedure. The POPDI is a six-item measure from the PFDI-20 which measures 6 different pelvic organ prolapse symptoms and degree of bother. The scale exists from 0-100 (0=no symptoms, 100=worse symptoms).
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Coloplast, Inc. Restorelle Y Mesh | Coloplast, Inc. Restorelle Dual Flat Mesh
Number analyzed (Participants) | 20 | 24
score on a scale | -32.5 (24.1) | -40.7 (26.9)

4. Secondary Outcome: Postoperative Mean Difference CRADI at 24 Months
Description: Mean difference between baseline (pre-procedure) and 24-months post-procedure. The CRADI is a eight-item measure from the PFDI-20 which measures 8 different pelvic organ prolapse symptoms and degree of bother. The scale exists from 0-100 (0=no symptoms, 100=worse symptoms).
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Coloplast, Inc. Restorelle Y Mesh | Coloplast, Inc. Restorelle Dual Flat Mesh
Number analyzed (Participants) | 20 | 24
score on a scale | -24.2 (20.6) | -20.2 (16.1)

5. Secondary Outcome: Postoperative Mean Difference UDI at 24 Months
Description: Mean difference between baseline (pre-procedure) and 24-months post-procedure. The UDI is a six-item measure from the PFDI-20 which measures 6 different pelvic organ prolapse symptoms and degree of bother. The scale exists from 0-100 (0=no symptoms, 100=worse symptoms).
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Coloplast, Inc. Restorelle Y Mesh | Coloplast, Inc. Restorelle Dual Flat Mesh
Number analyzed (Participants) | 20 | 24
score on a scale | -39.0 (27.0) | -33.2 (18.9)

6. Secondary Outcome: Postoperative Subjective Recurrence at 24 Months
Description: Subjective Recurrence was defined as patients who complained of vaginal bulge symptoms (Question #3 on the PFDI-20).
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Coloplast, Inc. Restorelle Y Mesh | Coloplast, Inc. Restorelle Dual Flat Mesh
Number analyzed (Participants) | 20 | 24
Participants | 2 | 2

7. Secondary Outcome: Postoperative Objective Recurrence at 24 Months
Description: Objective Recurrence
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Coloplast, Inc. Restorelle Y Mesh | Coloplast, Inc. Restorelle Dual Flat Mesh
Number analyzed (Participants) | 20 | 24
Participants | 5 | 4

8. Secondary Outcome: Reported Mesh Erosion at 24 Months
Description: Mesh Erosion was defined as presence of eroded mesh in the vagina on examination postoperatively up to 24-months after surgery.
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Coloplast, Inc. Restorelle Y Mesh | Coloplast, Inc. Restorelle Dual Flat Mesh
Number analyzed (Participants) | 20 | 24
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected up to 6 weeks after index surgery
Arm/Group | Coloplast, Inc. Restorelle Y Mesh | Coloplast, Inc. Restorelle Dual Flat Mesh
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/29
Other Adverse Events (participants affected / at risk) | 0/30 | 0/29

LIMITATIONS AND CAVEATS:
The biggest limitation in this study was lost to follow-up; however, this limitation was mitigated apriori by considering potential lost to follow-up in our power analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-08-26): https://cdn.clinicaltrials.gov/large-docs/87/NCT02156687/Prot_SAP_000.pdf